CLINICAL TRIAL: NCT00301574
Title: Placebo-Controlled, Double-Blind Study of Galantamine (R113675) in the Treatment of Alzheimer's Disease.
Brief Title: An Efficacy and Safety Study of Galantamine for the Treatment of Patients With Alzheimer's Disease.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR003301
Record Dates: First submitted 2006-03-10; First posted 2006-03-13 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2011-01

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer's disease; Cognitive dysfunction
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction | interventions — Galantamine

INTERVENTIONS:
Drug: galantamine

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of two fixed doses (16mg/day and 24mg/day) of galantamine (a drug for treating dementia) versus placebo for the treatment of patients with Alzheimer's disease, and to investigate the dose-response.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, parallel-group study to evaluate the efficacy and safety of two fixed doses of galantamine (16 and 24 milligrams per day [mg/day]) in patients with Alzheimer's disease, and to investigate the dose-response. The study consists of a 4-week screening period during which all patients will receive placebo, and a 22-week double-blind treatment period during which patients will receive placebo, galantamine 16 mg/day, or galantamine 24 mg/day. For patients receiving galantamine treatment, the starting dose is 8 mg/day and increases at 4-week intervals in increments of 8 mg/day. The primary measures of effectiveness are the change from baseline to the end of the study (week 22) in the Alzheimer's Disease Assessment Scale - Japan cognitive subscale (ADAS-J cog) and the Clinician's Interview-Based Impression of Change plus - Japan (CIBIC plus-J). Safety assessments include the incidence of adverse events, clinical laboratory tests, vital signs, electrocardiograms (ECGs), and physical examination findings. The study hypothesis is that galantamine will be more effective in the treatment of Alzheimer's disease than placebo. Study drug taken orally twice a day. 4-week screening period: All patients receive placebo. 22-week treatment period: Patients receive placebo, galantamine 16 mg/day, or 24 mg/day. For galantamine treatment, the starting dose is 8 mg/day and increases at 4-week intervals in increments of 8 mg/day.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients with a diagnosis of Alzheimer's disease according to the National Institute of Neurological and Communicative Disorders and the Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria
* having a Mini-Mental Status Examination (MMSE) score of 10 - 22 inclusive
* having an Alzheimer's Disease Assessment Scale - Japan cognitive subscale (ADAS-J cog) score of at least 18
* exhibiting an onset and progression of cognitive dysfunction during at least 6 months prior to the screening period

Exclusion Criteria:

* Patients with neurodegenerative diseases other than Alzheimer's disease, such as Lewy bodies disease, (dementia due to tiny round structures made of proteins that develop within nerve cells in the brain), Parkinsonism, etc
* Patients with cognitive dysfunction due to cerebral damage resulting from a lack of oxygen, a brain injury, etc
* Patients with multi-infarct dementia (brought on by a series of strokes) or active cerebrovascular disease
* Patients with clinically significant cardiovascular disease
* Patients currently taking drugs such as a cholinesterase inhibitors, which improve cerebral circulation/metabolism

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 398 (Actual)
Dates: Start 2001-04; Study Completion 2004-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline to the end of the study in the Alzheimer's Disease Assessment Scale - Japan cognitive subscale (ADAS-J cog) and the Clinician's Interview-Based Impression of Change plus - Japan (CIBIC plus-J)

SECONDARY OUTCOMES:
Change from baseline to the end of the study in CIBIC plus-J subscales (Disability Assessment for Dementia [DAD], Behavioral Pathology in Alzheimer's Disease Rating Scale [Behave-AD], the Mental Function Impairment Scale [MENFIS ]).

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K. Clinical Trial, Study Director — Janssen Pharmaceutical K.K.

REFERENCES:
- See also: An Efficacy and Safety Study of Galantamine in Patients with Alzheimer's Disease. — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=403&filename=CR003301_CSR.pdf